CLINICAL TRIAL: NCT03189017
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Trial in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ICP-022 Following Single and Multiple Escalating Dose
Brief Title: A Phase I Study of ICP-022 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innocare Pharma Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-001
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2018-07

CONDITIONS: Systemic Lupus Erythematosus; Rheumatoid Arthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICP-022 (Experimental): There are 5 cohorts in the Part 1 phase of the trial. Three quarters of subjects will be randomized to receive ICP-022 in a double-blind fashion. Five dose levels will be evaluated; dose escalation steps may be modified based on the safety from the previous dose. Cohort 4 will return on Day 8 and receive a single dose of ICP-022 under fed conditions.
  In Part 2 phase of the trial,three quarters of subjects will be randomized to receive the ICP-022 in a double-blind fashion in 3 cohorts. ICP-022 will be administered once a day for 14 consecutive days.
  Interventions: Drug: ICP-022
- Placebos (Placebo Comparator): In part 1 phase of the trial, one quarter of subjects will be randomized to receive placebo in a double-blind fashion. Cohort 4 will return on Day 8 and receive a single dose of placebo under fed conditions.
  In Part 2 phase of the trial,one quarter of subjects will be randomized to receive placebo in a double-blind fashion. Placebo will be administered once a day for 14 consecutive days.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: ICP-022 — The drug product is a white, round, uncoated tablet.
  Arms: ICP-022
Drug: Placebos — The placebo is a white, round, uncoated tablet.
  Arms: Placebos

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled, dose escalation study in healthy subjects to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ICP-022 following oral single and multiple escalating dose administration.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, dose escalation, placebo-controlled, first-in-humans phase 1 study to investigate the safety and tolerability of single and multiple escalating doses of ICP-022 in healthy volunteers. 40 healthy male participants (aged between 18 and 55 years of age inclusive) will be enrolled into Part 1 (single escalating dose administration) of this study, and additional 24 male subjects will be enrolled in Part 2 (multiple escalating dose administration). Part 1a consists of 5 cohorts of 8 participants each, while Part 2 includes 3 cohorts of 8 participants each.

Part 1a consists a treatment period with single oral dosing, and a safety follow-up to 7 days after dosing. Cohort 4 of Part 1a will return on Day 8 to repeat the study under fed condition in Part 1b.

Part 2 consists a treatment period with multiple dosing (once per day for 14 consecutive days), and a safety follow-up until 28 days after dosing. All subjects will receive either ICP-022 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects age ≥18 and ≤55 years
* Body mass index ≥19 and ≤31 kg/m2, with minimum body weight of 50kg
* No clinically significant findings in the medical history and physical examination, especially with regard to the respiratory, heart, immune system, pancreas, liver, bile and gastrointestinal systems
* No clinically significant laboratory values and urinalysis, unless the investigator considers any abnormality to be clinically irrelevant;
* Subjects with a partner of child-bearing potential must be willing to use an approved form of contraception with a failure rate of <1%. Subjects must be willing to use a condom during sexual intercourse whether or not their partner is of child-bearing potential from screening until 90 days after their final study visit.
* Normal electrocardiogram (ECG), blood pressure, and heart rate, unless the investigator considers any abnormality to be clinically irrelevant
* Informed consent must be obtained in writing for all subjects personally at enrollment

Exclusion Criteria:

* Subjects with medically important events
* Having 1st degree relative with coronary heart disease at age <60
* Using of prescription drugs including but not limited to those known to interfere with metabolism of drugs within 30 days prior to dosing
* Exposure to any other medication, including over-the-counter medications, herbal remedies and vitamins for at least 14 days before randomization (except paracetamol
* Participation in another study with any investigational drug in 30 days or five half-lives (whichever is longer) preceding the study
* Current smoker, defined as more than 10 cigarettes or equivalent per day before the beginning of the study (participants currently smoking ≤10 cigarettes daily and able to completely stop smoking during the study from screening until follow-up are eligible)
* Symptoms of a clinically significant illness in the 3 months before the study
* Presence or sequelae of respiratory, gastrointestinal, immune system, heart, liver or kidney disease, including asymptomatic unconjugated hyperbilirubinemia or asthma, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease
* Hemorrhoids or anal diseases with regular or recent presence of blood in feces
* History of immediate hypersensitivity to any medications or any food allergy, and acute phase of allergic rhinitis in the previous 2 weeks before randomization
* Blood or plasma donation of more than 500 mL during the previous 2 months before randomization and/or more than 50 mL in the 2 weeks prior to screening, or plan to donate any additional blood for 12 weeks after completing the study
* Subjects with a positive quantiFERON® test at screening or within 6 months prior to Day 1
* Positive test for human immunodeficiency virus (HIV)
* Positive test for hepatitis B (surface antigens HBs), or C (antibody HCs), unless caused by immunization
* Positive urine drug screen within 1 year before randomization
* Positive alcohol screen or active alcoholism
* Mental condition rendering the subject incapable to understand the nature, scope, and possible consequences of the study
* Subject has difficulty swallowing or is unable to swallow a tablet
* Unlikely to comply with the clinical study protocol eg, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study
* Investigator, or any sub-investigator, research assistant, pharmacist, study coordinator, other staff directly involved in the conduct of the protocol, or first degree relative thereof
* Subject requires anticoagulation treatment in the past 30 days
* Subject with anemia of any kind
* Subject with pancreatic abnormality of any kind, or elevated Lipase or Amylase >ULN

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | up to 28 days
  Number of participants with treatment-related adverse events will be collected and the percentage of AE of different grades will be assessed.

SECONDARY OUTCOMES:
Maximum plasma drug concentrations (Cmax) | up to 16 days
  Individual plasma concentrations of ICP-022 will be measured and Cmax will be calculated with noncompartmental analysis using WinNonlin.
Time of maximum plasma drug concentrations (Tmax) | up to 16 days
  Time of maximum plasma drug concentrations (Tmax) of ICP-022 will be recorded.
Area under the concentration time curve up to the time "t" (AUC(0-t)) | up to 16 days
  Area under the concentration time curve up to the time "t" (AUC(0-t)) of ICP-022 will be measured and calculated with noncompartmental analysis using WinNonlin.
Area under the concentration time curve up to the last data point above LOQ (AUC(last)) | up to 16 days
  Area under the concentration time curve up to the last data point above LOQ (AUC(last)) of ICP-022 will be measured and calculated with noncompartmental analysis using WinNonlin.
Apparent half-life for designated elimination phases (t½) | up to 16 days
  Apparent half-life for designated elimination phases (t½) of ICP-022 will be measured and calculated with noncompartmental analysis using WinNonlin.
Percent target occupancy | up to 16 days
  PBMC from individual subject before and after dosing will be collected and the target occupancy will be determined by ELISA. The percent of target occupancy will be compared descritively.

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, Principal Investigator — CMAX
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi J, Kim ST, Craft J. The pathogenesis of systemic lupus erythematosus-an update. Curr Opin Immunol. 2012 Dec;24(6):651-7. doi: 10.1016/j.coi.2012.10.004. Epub 2012 Nov 3. PMID 23131610
- [Background] Holroyd CR, Edwards CJ. The effects of hormone replacement therapy on autoimmune disease: rheumatoid arthritis and systemic lupus erythematosus. Climacteric. 2009 Oct;12(5):378-86. doi: 10.1080/13697130903025449. PMID 19591008
- [Background] Sanz I, Lee FE. B cells as therapeutic targets in SLE. Nat Rev Rheumatol. 2010 Jun;6(6):326-37. doi: 10.1038/nrrheum.2010.68. PMID 20520647
- [Background] Garcia A, De Sanctis JB. A Review of Clinical Trials of Belimumab in the Management of Systemic Lupus Erythematosus. Curr Pharm Des. 2016;22(41):6306-6312. doi: 10.2174/1381612822666160831103254. PMID 27587201
- [Background] Rovin BH, Furie R, Latinis K, Looney RJ, Fervenza FC, Sanchez-Guerrero J, Maciuca R, Zhang D, Garg JP, Brunetta P, Appel G; LUNAR Investigator Group. Efficacy and safety of rituximab in patients with active proliferative lupus nephritis: the Lupus Nephritis Assessment with Rituximab study. Arthritis Rheum. 2012 Apr;64(4):1215-26. doi: 10.1002/art.34359. Epub 2012 Jan 9. PMID 22231479
- [Background] Harandi A, Zaidi AS, Stocker AM, Laber DA. Clinical Efficacy and Toxicity of Anti-EGFR Therapy in Common Cancers. J Oncol. 2009;2009:567486. doi: 10.1155/2009/567486. Epub 2009 May 6. PMID 19424511
- See also: The Association of the British Pharmaceutical Industry (ABPI) represents innovative research-based biopharmaceutical companies, large, medium and small, leading an exciting new era of biosciences in the UK. — http://www.abpi.org.uk
- See also: AMH Online is the Australian Medicines Handbook for desktops, laptops, tablets and smartphones with internet access. — http://amhonline-amh-net-au.salus.idm.oclc.org